CLINICAL TRIAL: NCT00506766
Title: Promoting Self Care to Prevent Urinary Incontinence (UI): A Four-Year Follow-up
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01NR007618-02 (NIH)
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Urinary Incontinence; Bladder Control
Keywords: Urinary Incontinence; Self efficacy; Pelvic floor muscle training; Bladder training
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Bladder Health Class consisting of 6 weekly group sessions — 1 time
Behavioral: Practice PFMT and BT — As needed for 4 years
Behavioral: Clinic examination for pelvic muscle function — 1/year for 4 years
Behavioral: Record keeping in 3-day voiding diary — Every 6 months for 4 years

SUMMARY:
This study examined whether self-efficacy promoted adherence to Pelvic Floor Muscle Training (PFMT) and Bladder Training (BT) in women aged 55 and older.

DETAILED DESCRIPTION:
The study was designed to determine the capacity of self-efficacy to predict maintenance of the practices of PFMT and BT. Women in the treatment arm of the RCT attended a Bladder Health Class (PFMT & BT) to prevent UI. The class content emphasized self-efficacy. At 3-months post intervention the self-efficacy of participants was measured; these results were collected to analyze for predictive capacity of training adherence. For four years participants in both the treatment and control (no class) arms were followed with both questionnaires and 3-day bladder diaries (2/year) and clinic evaluations of (1/year). In addition, qualitative analyses of the narratives of Bladder Health Class participants identified individual attitudes and strategies that either facilitated or deterred adherence.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 55 years or older who report 5 or fewer episodes of UI / year, no prior treatment for UI, no neurological disease, no difficulties performing activities of daily living

Exclusion Criteria:

* Less than 55 years old, UI episodes greater that 5 per year, score of less than 24 on Mini Mental Status Examination

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2000-09; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Adherence to PMFT and BT (self efficacy) were measured through questionnaires and 3-day voiding diaries. | Every 6 months for 4 years

SECONDARY OUTCOMES:
Adherence to PMFT and BT (self efficacy) were measured through questionnaires and days of urinary incontinence per 3-day voiding diary | Every 6 months for 4 years
Digital measurement during clinical examination of pelvic muscle function (pressure and displacement). | 1/year for four years
Paper towel bladder test | 1/year for four years
Survey questions (open ended and forced choice) about strategies women use to incorporate PFMT and BT into their lives | 1 time

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn M Sampselle, PhD,RNC,FAAN, Principal Investigator — University of Michigan School of Nursing; Sandra H Hines, PhD, RNC, Study Director — University of Michigan School of Nursing
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Hines SH, Seng JS, Messer KL, Raghunathan TE, Diokno AC, Sampselle CM. Adherence to a behavioral program to prevent incontinence. West J Nurs Res. 2007 Feb;29(1):36-56; discussion 57-64. doi: 10.1177/0193945906293793. PMID 17228060
- [Result] Messer KL, Herzog AR, Seng JS, Sampselle CM, Diokno AC, Raghunathan TE, Hines SH. Evaluation of a mass mailing recruitment strategy to obtain a community sample of women for a clinical trial of an incontinence prevention intervention. Int Urol Nephrol. 2006;38(2):255-61. doi: 10.1007/s11255-006-0018-1. PMID 16868693
- [Result] Sampselle CM, Messer KL, Seng JS, Raghunathan TE, Hines SH, Diokno AC. Learning outcomes of a group behavioral modification program to prevent urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2005 Nov-Dec;16(6):441-6. doi: 10.1007/s00192-005-1284-7. Epub 2005 Mar 15. PMID 16237512
- [Result] Sampselle CM, Palmer MH, Boyington AR, O'Dell KK, Wooldridge L. Prevention of urinary incontinence in adults: population-based strategies. Nurs Res. 2004 Nov-Dec;53(6 Suppl):S61-7. doi: 10.1097/00006199-200411006-00010. PMID 15586150
- [Result] Sampselle CM. Teaching women to use a voiding diary. Am J Nurs. 2003 Nov;103(11):62-4. doi: 10.1097/00000446-200311000-00031. No abstract available. PMID 14625427
- [Result] Diokno AC, Sampselle CM, Herzog AR, Raghunathan TE, Hines S, Messer K, Karl C, Leite MC. Prevention of urinary incontinence by behavioral modification program: a randomized, controlled trial among older women in the community. J Urol. 2004 Mar;171(3):1165-71. doi: 10.1097/01.ju.0000111503.73803.c2. PMID 14767293
- [Result] Sampselle CM. Behavioral interventions in young and middle-age women: simple interventions to combat a complex problem. Am J Nurs. 2003 Mar;Suppl:9-19. doi: 10.1097/00000446-200303001-00003. No abstract available. PMID 12612489
- [Result] Longworth, J, Davila, Y, Sampselle, CM. (2003) La perdida de orina: Hispanic women's experience of urinary incontinence. Hispanic Health Care International (The official Journal of the National Association of Hispanic Nurses), Vol. 2(1), 13-21.
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598